CLINICAL TRIAL: NCT05284487
Title: Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate Safety and Efficacy of Jalosome® Soothing Gel in the Prevention and Treatment of Radiation-induced Dermatitis in Patients With Head and Neck Cancer.
Brief Title: Clinical Trial to Evaluate Safety and Efficacy of Jalosome® Soothing Gel.
Acronym: JALOSOME-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Welcare Industries SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JALOSOME-01
Record Dates: First submitted 2022-02-04; First posted 2022-03-17 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2023-03

CONDITIONS: Radiation-induced Dermatitis
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Jalosome® Soothing gel (Active Comparator): Jalosome® soothing gel ((L-Acetyl Carnitine chloridrate, Allantoin, Hydrogenated phosphatidylcholine, Sodium Hyaluronate) will be applied to the irradiated area two times daily (morning after RT and evening). The first application will start in the morning after the first RT session and will continue up to two weeks after completion of RT.
  Visit 1: Screening (days -7 to 0) Visit 2: Randomization and start of RT (day 1) Visit 3 -Visit 9/10: RT treatment Last visit: 2 weeks after last RT
  Interventions: Device: Jalosome® soothing gel
- Group 2: Placebo (Placebo Comparator): Placebo will be applied to the irradiated area two times daily (morning after RT and evening). The first application will start in the morning after the first RT session and will continue up to two weeks after completion of RT.
  Visit 1: Screening (days -7 to 0) Visit 2: Randomization and start of RT (day 1) Visit 3 -Visit 9/10: RT treatment Last visit: 2 weeks after last RT
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Jalosome® soothing gel — Jalosome® Soothing gel is a phospholipid based vesicular system based on hyaluronic acid (HA). HA supports the process of formation of extracellular matrix and collagen synthesis by fibroblasts, favoring the formation of a well-vascularized granulation tissue and thus accelerating the healing process. Jalosome® Soothing gel contains other active ingredients: Acetyl-L-carnitine which plays an important role as shuttle for energy production and is involved in cellular metabolism. It is an effective cytoprotective, anti-inflammatory, neuroprotective, metal chelator, anti-apoptotic and anti-oxidant agent. Allantoin is a key constituent of comfrey (Symphytum officinale L), it has moisturizing and keratolytic effect, increasing the water content of the extracellular matrix and enhancing desquamation of upper layers of dead skin cells. Hydrogenated phosphatidylcholine is a permeation enhancers, which increases the solubilization of active ingredients, improving their skin permeation ability.
  Arms: Group 1: Jalosome® Soothing gel
Device: Placebo — The placebo does not contain the active ingredients of Jalosome, only the co-formulants.
  Arms: Group 2: Placebo

SUMMARY:
Primary objective

- To investigate the effectiveness of Jalosome® compared with placebo in the prevention and treatment of RID in patients with HNC undergoing RT.

Secondary objectives:

* To investigate the effectiveness of Jalosome® in reducing the maximum severity of RID compared with placebo.
* To investigate the effect of Jalosome®, compared with placebo, on patients' quality of life.
* To investigate safety and tolerability of Jalosome®.
* To investigate patient's compliance to Jalosome® treatment.
* To investigate patient's global satisfaction with Jalosome® treatment.

DETAILED DESCRIPTION:
Primary endpoint:

* Mean time difference in development of G2 RID (according to CTCA) between Jalosome® and placebo arms. A median difference of at least 7 days is considered of clinical significance.

  • Secondary endpoints:
* Proportion of subjects without G2 RID at the end of RT, in the Jalosome® and placebo arms.
* Proportion of subjects without G2 RID at different timepoints (week 5, week 6 and two weeks after the last radiation) in the Jalosome® and placebo arms.
* Worst skin toxicity during treatment and up to 2 weeks after the last radiation, according to CTCAE, in the Jalosome® and placebo arms.
* RID grade (mean and worst) on the RISRAS scale, assessed weekly, in the Jalosome® and placebo arms.
* Mean and worst score of PRO-Skindex-16 questionnaire performed weekly, in the Jalosome® and placebo arms.
* Mean pain measured by the 11-point NRS of the Brief Pain Inventory (BPI), as reported in patients' diary (daily) and assessed during visits (weekly), in the Jalosome® and placebo arms.
* Patient's compliance to Jalosome® treatment.
* Patient's global satisfaction with Jalosome® treatment.
* Jalosome® overall safety and tolerability.

Study design:

Monocentric, randomized, double-blind, placebo controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subject aged ≥18 years old.
* Performance status 0-1.
* Diagnosis of HNC (epithelial carcinoma of oropharynx, nasopharynx, larynx, hypopharynx, paranasal sinuses or salivary glands).
* Postoperative or curative RT (total radiation dose of at least 60 Gy), with or without concurrent chemotherapy.
* Willingness and ability to give informed consent and comply with study procedures.

Exclusion Criteria:

* Pregnant or lactating women.
* Previous RT on the head and neck area.
* Planned to receive concurrent cetuximab.
* Cutaneous and/or connective diseases (i.e. lupus erythematosus or scleroderma).
* Systemic diseases known to delay the skin healing process, such as diabetes mellitus or severe renal failure.
* Use of a tissue-equivalent bolus.
* Use of over-the-counter topical medications containing steroids.
* Presence of rashes or unhealed wounds in the radiation field.
* Recent sun exposure (<1 month).
* Mental conditions that could adversely affect subject's adherence to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Time to development of G2 RID | 9 weeks
  Mean number of days in development of G2 RID (according to CTCA), in the Jalosome® and placebo arms.

SECONDARY OUTCOMES:
Subjects without G2 RID at the end of RT | 9 weeks
  Number and percentage of subjects without G2 RID at the end of RT, in the Jalosome® and placebo arms..
Subjects without G2 RID at different timepoints | 9 weeks
  Number and percentage of subjects without G2 RID at different timepoints (week 5, week 6 and two weeks after the last radiation) in the Jalosome® and placebo arms.
Worst skin toxicity | 9 weeks
  Number and percentage of subjects with worst skin toxicity G3, G2 and G1 RID according to CTCAE v.4.0, during treatment and up to 2 weeks after the last administration of RT, in the Jalosome® and placebo arms.
RID grade on the RISRAS | 9 weeks
  Mean RID grade on the Radiation-Induced Skin Reaction Assessment Scale scale (RISRAS), assessed weekly, in the Jalosome® and placebo arms.
  RISRAS score varies from 0 to 36, where 0 is normal skin/no symptoms at all and 36 is the worst conditions in terms of erythema-Dry desquamation - Moist desquamation - necrosis of derma (14 points) and very severe symptoms (12 points).
PRO-Skindex-16 questionnaire score | 9 weeks
  Mean score of each item (16 items) of PRO-Skindex-16 questionnaire performed weekly, in the Jalosome® and placebo arms. Each item is about skin discomfort, ancd the scores vary from 0 (no discomfort) to 6 (full discomfort).
Pain measured by NRS | 9 weeks
  Mean pain measured by the 11-point Numeric rating scale (NRS) of the Brief Pain Inventory (BPI), as reported in patients' diary (daily) and assessed during visits (weekly), in the Jalosome® and placebo arms.
  NRS score varies from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Compliance | 9 weeks
  Number and percentage of patients with compliance to Jalosome® treatment ≥80%.
Adverse events | 9 weeks
  Number and percentage of adverse events by grade, according to the CTCAE v.4.0, and relationship with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Alessandro Iacovelli, Principal Investigator — Fondazione IRCCS ISTITUTO NAZIONALE TUMORI
Locations (1):
- IRCCS, Milan, Italy